CLINICAL TRIAL: NCT01254539
Title: Phase I/II Clinical Trial on The Use of Autologous Bone Marrow Stem Cells in Amyotrophic Lateral Sclerosis (Extension CMN/ELA)
Brief Title: Clinical Trial on The Use of Autologous Bone Marrow Stem Cells in Amyotrophic Lateral Sclerosis (Extension CMN/ELA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Universitario Virgen de la Arrixaca (Other); Hospital General Universitario Morales Meseguer (Other); Diógenes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Extension CMN/ELA; 2006-003096-12 (EudraCT Number); EC07/90762 (Other: ISCIII)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2015-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Bone marrow; Stem cells; Autologous; Safety
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Laminectomy; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autologous bone marrow stem cells intraspinal transplantation (Experimental): T3-T4 laminectomy and bone marrow ficoll separated mononuclear autologous cells intraspinal transplantation
  Interventions: Procedure: Laminectomy and bone marrow stem cells transplantation
- Intrathecal infusion of autologous bone marrow stem cells (Experimental): Patients were drawn 2 ml of cerebrospinal fluid and infused 2 ml (two 1 ml syringes) of Autologous Stem Cells.
  Interventions: Procedure: Intrathecal infusion of autologous bone marrow stem cells
- Intrathecal infusion of placebo (saline solution). (Placebo Comparator): Patients were infused 2 ml of saline solution
  Interventions: Procedure: Intrathecal infusion of placebo (saline solution).

INTERVENTIONS:
Procedure: Laminectomy and bone marrow stem cells transplantation — Autologous bone marrow cells collection under sedation. Sixty ml are obtained and processed through a ficoll gradient.
  T3-T4 laminectomy and bone marrow ficoll separated mononuclear autologous cells intraspinal transplantation
  Arms: Autologous bone marrow stem cells intraspinal transplantation
Procedure: Intrathecal infusion of autologous bone marrow stem cells — Autologous bone marrow cells collection under sedation. Sixty ml are obtained and processed through a ficoll gradient.
  Patients were drawn 2 ml of cerebrospinal fluid and infused 2 ml (two 1 ml syringes) of Autologous Stem Cells.
  Arms: Intrathecal infusion of autologous bone marrow stem cells
Procedure: Intrathecal infusion of placebo (saline solution). — Patients were infused 2 ml of saline solution
  Arms: Intrathecal infusion of placebo (saline solution).

SUMMARY:
The purpose of this clinical trial is to assess the feasibility and the security of the intraspinal and intrathecal infusion of autologous bone marrow stem cells for the treatment of Amyotrophic Lateral Sclerosis patients.

DETAILED DESCRIPTION:
Patients with Amyotrophic Lateral Sclerosis (ALS) typically endure a progressive paralysis due to the continued loss of motoneurons that leads them to death in less than 5 years. No treatment has changed its natural history. Intraspinal injections of bone marrow mononuclear cells (MNC) have been able to ameliorate the course of ALS in murine models, acting as pumps of trophic factors that keep the motoneurons functional. Moreover, the clinical trial (Study NCT00855400 on www.ClinicalTrials.gov) conducted by our research group to determine the safety and efficacy of Autologous Stem Cell transplantation in Amyotrophic Lateral Sclerosis in humans, found that this procedure is feasible and safe. Continuing with that study, we have designed a phase I/II clinical trial to check the feasibility of the intraspinal and intrathecal infusion of autologous bone marrow stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose established following the World Federation of Neurology criteria
* More than 6 and less than 36 months of evolution of the disease
* Medullar onset of the disease
* More than 18 and less than 70 years old
* Forced Vital Capacity ≥ 50%
* Total time of oxygen saturation <90% inferior to 5% of the sleeping time
* Signed informed consent

Exclusion Criteria:

* Neurological or psychiatric concomitant disease
* Need of parenteral or enteral nutrition through percutaneous endoscopic gastrostomy or nasogastric tube
* Concomitant systemic disease
* Treatment with corticosteroids, immunoglobulins or immunosuppressors during the last 12 months
* Inclusion in other clinical trials
* Unability to understand the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-10; Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | Every 3 months

SECONDARY OUTCOMES:
Neurological variables: The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALS-FRS), Medical Research Council (MRC) and Norris scales | Every 3 months
Absence of adverse events | Every week / month depending on the study phase
Neurophysiological variables: Electromyography, polysomnography, evoked potentials | Every 3 months
Neuroradiological variables: Spinal Magnetic Resonance Imaging (MRI) | Every 3 months
Respiratory variables: Maximal inspiratory pressure (PIM), Maximal expiratory pressure (PEM), sniff nasal, oxymetry. | Every 3 months
Psychological variables: Health Questionnaire (EuroQol-5D), The Profile of Mood States (POMS) | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose María Moraleda Jiménez, M.D. PhD., Study Director — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain

REFERENCES:
- See also: Spanish Cell Therapy Network — http://red-tercel.com/
- See also: Amyotrophic Lateral Sclerosis — http://www.ncbi.nlm.nih.gov/mesh/68000690